CLINICAL TRIAL: NCT06301035
Title: Comparison of Asymmetric High-flow Nasal Cannula (HFNC) and Standard HFNC in Post Extubation High-risk Group: A Prospective, Single-center, Open-labeled, Randomized Controlled Pilot Study
Brief Title: Asymmetric High-flow Nasal Cannula (HFNC) vs Standard HFNC for Post Extubation High-risk Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Chi Ryang Chung, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-01-012
Record Dates: First submitted 2024-01-22; First posted 2024-03-08 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Failure
Keywords: High flow nasal cannula; Electrial impedance tomography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asymmetric HFNC (Experimental): Asymmetric HFNC
  Interventions: Device: Asymmetric High flow nasal cannula
- Standard HFNC (Active Comparator): Standard HFNC
  Interventions: Device: Standard(symmetric) High flow nasal cannula

INTERVENTIONS:
Device: Asymmetric High flow nasal cannula — * Both the test group and the control group apply high flow oxygen therapy for at least 24 hours from the time of initial excretion (0h), and only the nasal interface is applied differently depending on the allocation group.
  * The initial flow rate setting is 10 L/min, and it can be adjusted up to 50 L/min within the range where the subject does not experience discomfort. Except for cases where the patient complains of being hot, the initial temperature setting is 37°C, and the inhaled oxygen concentration (FiO2) may be adjusted to a target of 93% or more of peripheral oxygen saturation (SpO2) in the range of 21 to 100%.
  * After 24 hours, high flow oxygen therapy is discontinued and conventional oxygen therapy can be applied if necessary.
  Arms: Asymmetric HFNC
Device: Standard(symmetric) High flow nasal cannula — * Both the test group and the control group apply high flow oxygen therapy for at least 24 hours from the time of initial excretion (0h), and only the nasal interface is applied differently depending on the allocation group.
  * The initial flow rate setting is 10 L/min, and it can be adjusted up to 50 L/min within the range where the subject does not experience discomfort. Except for cases where the patient complains of being hot, the initial temperature setting is 37°C, and the inhaled oxygen concentration (FiO2) may be adjusted to a target of 93% or more of peripheral oxygen saturation (SpO2) in the range of 21 to 100%.
  * After 24 hours, high flow oxygen therapy is discontinued and conventional oxygen therapy can be applied if necessary.
  Arms: Standard HFNC

SUMMARY:
Background The exacerbation of respiratory failure that occurs after endotracheal intubation often occurs in patients who have received mechanical ventilation therapy, and when it occurs, it emerges as an important issue to consider reintubation of endotracheal intubation. High-flow nasal cannula (HFNC) through nasal cannula is known to produce positive airway pressure and deliver a certain amount of oxygen, and recently reported clinical studies have demonstrated the effect of lowering the risk of reintubation after endotracheal intubation, which is recommended for use in recent clinical practice guidelines. However, in patients at high risk of intubation failure, the combination of high-flow oxygen therapy and non-invasive positive-pressure ventilation therapy rather than the application of high-flow oxygen therapy alone through nasal cannula is helpful in reducing the rate of reintubation of endotracheal intubation. However, an alternative to non-invasive positive-pressure ventilation therapy is needed as there is a possibility of complications such as aspiration pneumonia, maladaptation of the application device (mask), and discomfort, making it difficult to apply it in the field.

Recently, it has been reported that high flow oxygen therapy through an asymmetric nasal cannula forms sufficient positive pressure in terms of respiratory dynamics, which makes the patient feel comfortable and reduces work of breath. However, no clinical studies have yet compared physiological effects using this method in patients at high risk of extubation failure.

Goal The investigators would like to compare the physiological effects of high flow oxygen therapy through 'asymmetric nasal cannula' with high flow oxygen therapy through 'standard nasal cannula' in patients identified as high-risk groups for valvular failure.

Hypothesis 'Asymmetric nasal cannula' reduces work of breath compared to 'standard nasal cannula' in high-risk patients with valvular failure.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years of age or older
2. Patients who applied mechanical ventilation treatment for more than 24 hours before the excision
3. Patients who underwent endotracheal intubation rather than tracheal incision
4. Planned extubation after successful spontaneous breathing trial (SBT)
5. Reintubation High Risk Patients: If any of the following conditions are met

   1. Age > 65
   2. Acute Physiology and Chronic Health Evaluation(APACHE) II on the day of extubation > 12
   3. Body mass index (BMI) > 30 kg/m2
   4. Inability to deal with respiratory secretions

      * improper cough reflex
      * If at least three aspirations are required in the 8 hours prior to the discharge
   5. Difficult or long delay in mechanical ventilation

      * The first attempt to leave the mechanical ventilation failed
   6. Charlson Commercial Index (CCI) at least 2 categories of comorbidities
   7. Heart failure is the main indication of mechanical ventilation application
   8. Moderate to severe chronic obstructive pulmonary disease
   9. If there is a problem with airway openness (high risk of developing laryngeal edema)

      * a woman
      * Oral endotracheal intubation maintenance period of at least 3 days
      * Difficult to intubate endotracheally (difficult airway)
   10. Long-term mechanical ventilation application: When applied for more than 7 days

Exclusion Criteria:

1. a patient with a tracheostomy tube
2. Contraindicated application of nasal interfaces

   * a nasal disorder
3. Continuous positive pressure (CPAP) application contraindications

   * pneumothorax, blistering lung disease, head trauma, cranial facial surgery, airway foreign matter, unstable hemodynamics, etc
4. EIT application contraindications

   * Patients using implantable electronic medical devices (such as implantable defibrillators, pacemakers or spinal cord stimulators)
   * a patient with hyperhidrosis
   * a patient whose physical movements are not controlled
   * a pregnant woman
   * BMI 50 or higher

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate Oxygenation (ROX) Index | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  Changes in Respiratory Rate Oxygenation (ROX) Index after extubation
  4.88 ≤ ROX index ; Low Risk 3.85 ≤ ROX index < 4.88 ; Re-evaluate after 1-2 hours 3.85 > ROX index ; considerate about intubation

SECONDARY OUTCOMES:
The Lowest value of SpO2 within 24 hours after extubation | within 24 hours after extubation
  Gas exchange (blood gas analysis) - The Lowest value of SpO2 within 24 hours after extubation
PaO2/FiO2 | 30 minutes, 6 hours, 24 hours
  Gas exchange (blood gas analysis) - PaO2/FiO2
SpO2/FiO2 | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  Gas exchange (blood gas analysis) - SpO2/FiO2
changes of end-expiratory lung impedance, at each flow rate measured through Electrical Impedance tomography (EIT) | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  Pulmonary Dynamics (EIT) - changes of end-expiratory lung impedance, at each flow rate measured through Electrical Impedance tomography (EIT)
Changes in non-homogeneity indicators measured through EIT (changes in Global homeogeneity index) | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  Pulmonary Dynamics (EIT) - Changes in non-homogeneity indicators measured through EIT (changes in Global homeogeneity index)
Respiratory rate | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  respiratory capacity indicator - Respiratory rate
work of breath (Modified Borg Scale, MBS) | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  respiratory capacity indicator - work of breath (Modified Borg Scale, MBS)
  :The degree of work of breath is indicated by the patient himself/herself 0: Nothing at all 0.5: Very, very slight (just noticeable)
  1. Very slight
  2. Slight
  3. Moderate
  4. Somewhat severe 5,: Severe 6, 7: Very severe 8, 9: Very, very severe (almost maximal)
  10: Maximal
systolic blood pressure | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  hemodynamics - systolic blood pressure
mean arterial pressure | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  hemodynamics - mean arterial pressure
heart rate | 1 hour, 2 hours, 6 hours, 12 hours, 24 hours
  hemodynamics - heart rate
Rate of reintubation within 7 days | within 7 days after extubation
  clinical outcomes - Rate of reintubation within 7 days
Length of ICU stay | From date of ICU admission until the date of ICU discharge, assessed up to 2 years
  clinical outcomes - Length of ICU stay
Length of hospital stay | From date of hospital admission until the date of hospital discharge, assessed up to 2 years
  clinical outcomes - Length of hospital stay
ICU Mortality | From date of extubation until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 1 year
  clinical outcomes - ICU Mortality
Hospital Mortality | From date of extubation until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 1 year
  clinical outcomes - Hospital Mortality
28 Day Mortality | From date of extubation until the date of 28 Day or date of death from any cause, whichever came first, assessed up to 1 months
  clinical outcomes - 28 Day Mortality
90 Day Mortality | From date of extubation until the date of 90 Day or date of death from any cause, whichever came first, assessed up to 3 months
  clinical outcomes - 90 Day Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Background] Thille AW, Muller G, Gacouin A, Coudroy R, Decavele M, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Cabasson S, Rouze A, Vivier E, Le Meur A, Ricard JD, Razazi K, Barberet G, Lebert C, Ehrmann S, Sabatier C, Bourenne J, Pradel G, Bailly P, Terzi N, Dellamonica J, Lacave G, Danin PE, Nanadoumgar H, Gibelin A, Zanre L, Deye N, Demoule A, Maamar A, Nay MA, Robert R, Ragot S, Frat JP; HIGH-WEAN Study Group and the REVA Research Network. Effect of Postextubation High-Flow Nasal Oxygen With Noninvasive Ventilation vs High-Flow Nasal Oxygen Alone on Reintubation Among Patients at High Risk of Extubation Failure: A Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1465-1475. doi: 10.1001/jama.2019.14901. PMID 31577036
- [Background] Slobod D, Spinelli E, Crotti S, Lissoni A, Galazzi A, Grasselli G, Mauri T. Effects of an asymmetrical high flow nasal cannula interface in hypoxemic patients. Crit Care. 2023 Apr 18;27(1):145. doi: 10.1186/s13054-023-04441-6. PMID 37072854
- [Background] Tan D, Walline JH, Ling B, Xu Y, Sun J, Wang B, Shan X, Wang Y, Cao P, Zhu Q, Geng P, Xu J. High-flow nasal cannula oxygen therapy versus non-invasive ventilation for chronic obstructive pulmonary disease patients after extubation: a multicenter, randomized controlled trial. Crit Care. 2020 Aug 6;24(1):489. doi: 10.1186/s13054-020-03214-9. PMID 32762701
- [Background] Hernandez G, Paredes I, Moran F, Buj M, Colinas L, Rodriguez ML, Velasco A, Rodriguez P, Perez-Pedrero MJ, Suarez-Sipmann F, Canabal A, Cuena R, Blanch L, Roca O. Effect of postextubation noninvasive ventilation with active humidification vs high-flow nasal cannula on reintubation in patients at very high risk for extubation failure: a randomized trial. Intensive Care Med. 2022 Dec;48(12):1751-1759. doi: 10.1007/s00134-022-06919-3. Epub 2022 Nov 18. PMID 36400984
- [Background] Tatkov S, Rees M, Gulley A, van den Heuij LGT, Nilius G. Asymmetrical nasal high flow ventilation improves clearance of CO2 from the anatomical dead space and increases positive airway pressure. J Appl Physiol (1985). 2023 Feb 1;134(2):365-377. doi: 10.1152/japplphysiol.00692.2022. Epub 2023 Jan 12. PMID 36633864